CLINICAL TRIAL: NCT06199011
Title: Effect of Intraoperative Esketamine Infusion on Depressive Symptoms of Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Effect of Esketamine on Depressive Symptoms of Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy
Acronym: EDSOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Chunxia Huang, Associate Professor, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDSOP
Record Dates: First submitted 2023-12-14; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: Standardized general anesthesia (Active Comparator): The control group is standard of opioid anesthesia including reminfentanil and sufentanil. In addition to dexmedetomidine and transverse abdominal plane block, general anesthesia induction will be induced performed with sufentanil (0.5 μg kg-1), propofol (1.5 mg kg-1), and rocuronium (1 mg kg-1). General anesthesia was maintained with a continuous infusion of remifentanil (5-15 μg kg-1 h-1), cisatracurium (0.1-0.2 mg kg-1 h-1), dexmedetomidine (0.4 μg kg-1 h-1), and sevoflurane exposure guided by bispectral index. Dexmedetomidine administration and sevoflurane inhalation will be completed at 20 minutes before surgery finish. Propofol and remifentanil will be continuously infused till the end of surgery.
  Interventions: Drug: Opioid
- Intervention Group: A standardized non-opioid anesthesia (Experimental): Dexmedetomidine (0.5μg kg-1) and esketamine (0.25mg kg-1) was intravenously infused to provide sedation for the bilateral transverse abdominal plane block (0.33% ropivacaine and dexmedetomidine 1μg kg-1). General anesthesia was then induced with esketamine (0.25 mg kg-1 h-1), propofol (1.5 mg kg-1), and rocuronium (1 mg kg-1). Following endotracheal intubation, GA was maintained with a continuous infusion of esketamine (0.25 mg kg-1 h-1), cisatracurium (0.1-0.2 mg kg-1 h-1), dexmedetomidine (0.4 μg kg-1 h-1), and sevoflurane guided by bispectral index. The infusions of esketamine and dexmedetomidine, as well as sevoflurane inhalation will be finished at 20 minutes before surgery completion. Propofol will be continuously infused to maintain appropriate bispectral index.
  Interventions: Drug: Esketamine hydrochloride

INTERVENTIONS:
Drug: Esketamine hydrochloride — A standardized non-opioid anesthesia will be achieved by using continuous intraoperative infusion of esketamine.
  Arms: Intervention Group: A standardized non-opioid anesthesia
Drug: Opioid — A standardized opioid anesthesia will be achieved by using continuous intraoperative infusion of opioids.
  Arms: Control Group: Standardized general anesthesia

SUMMARY:
Esketamine, as a powerful analgesic intravenous anesthetic, has a rapid onset and elimination effect, does not inhibit spontaneous respiration, and can slightly stimulate the circulatory system. It has been confirmed that esketamine can effectively combat opioid related complications, especially life-threatening respiratory suppression. Thus becoming a new powerful perioperative analgesic drug. At the same time, esketamine has been licensed for the treatment of "resistant depression" and emergency treatment for patients in crisis states of depression. But the evidence for its safety and effectiveness is insufficient. We have designed a randomized controlled clinical trial to investigate the effect of an established general anesthesia strategy without opioids by using esketamine on postoperative depressive in obese patients undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
The bidirectional relationship between obesity and mood disorders is suggested supported by empirical evidence. Obesity increases the risk of depression, and depression predicts the developing of obesity. The associations between atypical depressive symptoms and obesity-related characteristics may consequent to sharing pathophysiologic characteristics in patients with major depressive disorders, such as genetics, and brain circuitries integrating homeostatic and mood regulatory responses.

Bariatric surgery is a remarkably effective and durable treatment for obesity, resulting in considerable weight loss, and reductions in the prevalence of type 2 diabetes mellitus, hypertension, dyslipidemia and sleep apnea at 5 years. Nearly 23-33% of patients undergoing bariatric surgery report a preoperative depression. Meanwhile, bariatric surgery is consistently associated with postoperative decreases in the prevalence of depression (8%-74% decrease) and the severity of depressive symptoms (40%-70% decrease) at 6-month, 12-month, 24-month. In 357 extremely obese patients with a mean BMI of 51.2 kg/m2, 45% of patients are identified as depression before gastric bypass surgery. And by 6-, 12-, 24-month follow-up, by using Beck Depression Inventory, clinically significant depressive symptoms are characterized to 12%, 13% and 18%, respectively. Compared with status prior to surgery, the prevalence of any Axis I psychiatric disorder for DSM-IV at 2 and 3 years after Roux-en-Y gastric bypass or laparoscopic adjustable gastric band surgery is significantly reduced from 30.2% to 16.8% and 18.4%.

Based on the HAMD assessments, we found that the incidence of depressive symptoms was 71.1% in 225 young obese patients (31.0 years-old) before laparoscopic sleeve gastrectomy. The depressive symptoms and severity were improved over time, particular in postoperative 3 months. However, depressive symptoms were still sustained in a proportion of obese patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥40kg/m2 or BMI>35 kg/m2 with an existing comorbidity
* scheduled for selective LSG
* American Society of Anesthesiologists physical status I-III
* HAMD>7
* with informed consent

Exclusion Criteria:

* Patients diagnosed with significant comorbidities, such as cardiopathy, chronic respiratory conditions, abnormal hepatic and/or renal function, coagulation dysfunction, major psychiatric or neurological disorders
* Patients allergy to esketamine or other drugs used in the study
* Patients are scheduled for/plan to have an additional surgery during the 3-month follow-up period
* Patients suffer from acute or chronic pain with analgesics, or take anticathartic, glucocorticoid medications
* Patients involved in another research study
* Patients will likely have problems, in the judgement of the investigator, with maintaining follow-up
* Any other reasons the investigator feels is relevant for excluding the patient
* lack of patient consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton depression Rating Scale | Before surgery and at the postoperative 3 months
  The 24-item version of the Hamilton Depression Scale (HAM-D) is used to assess the severity of depression. Each item is rated on the Likert scale, ranging from 0 to 4. The normal value is 0-7 points, the mild depression value is 8-20 points, the moderate depression symptom value is 21-35 points, and the severe depression value exceeds 35 points. The higher scores indicate the worse symptoms.

SECONDARY OUTCOMES:
Postoperative anxiety | In 3 months after surgery
  Postoperative anxiety
Hamilton Anxiety Rating Scale | Before surgery and at the postoperative 3 months
  Hamilton Anxiety Rating Scale (HAMA) will be used to assess anxiety. Total score ranges from 0 to 56, the higher the score is, the more serious the anxiety is.
Cognition | Before surgery and at the postoperative 3 months
  AVLT, Trail Making Tests, Stroop color and word test, word fluency, Digit span test will be used to evaluate the cognition.
The incidence of Postoperative nausea and vomiting | At 0-24 hours after surgery
  The incidence of Postoperative nausea and vomiting
Postoperative depressive symptoms | In 3 months after surgery
  Montgomery-Asberg Depression Rating Scale (MARDS) includes 10 items. The normal value is less than 12 points, the mild depression value is 12-22 points, the moderate depression symptom value is 22-30 points, and the severe depression value is 30-35 points, extreme severe depression value exceeds 35. The higher scores indicate the worse symptoms.
Postoperative pain | At 0-24 hours after surgery
  Postoperative incision pain and visceral pain will be assessed by VAS withing 0-10. The higher scores indicate the more pain.
Time to the first rescue analgesics | At 0-24 hours after surgery
  The time from extubation to the first rescue analgesics
Time to the first rescue antiemetics | At 0-24 hours after surgery
  The time from extubation to the first rescue antiemetics
Consumption of anesthetics | During the surgery
  Total usage of anesthetics during the surgery
Length of surgery | At the end of surgery
  From beginning to the end of surgery
Length of anesthesia | At the end of anesthesia
  From beginning to the end of anesthesia
QoR-15 | At 24 hours after surgery
  The QoR-15 is a convenient patient-reported tool, including 15 items of five domains (pain, comfort, physical independence, psychological support, and emotional state) with each item ranging from 0 to 10. Higher scores suggest better quality of recovery (0-89, poor recovery; 90-121, moderate recovery; 122-135, good recovery; 136-150, excellent recovery)
Adverse event rate | During postoperative 3 months
  The incidence of adverse events
BMI | Before surgery and at the postoperative 3 months
  Body mass index
Pittsburgh Sleep Quality Index | Before surgery and at the postoperative 3 months
  Pittsburgh Sleep Quality Index (PSQI) will be assessed the quality of sleep. The higher score means the lower quality of sleep.
Gastrointestinal Symptom Rating Scale | Before surgery and at the postoperative 3 months
  Gastrointestinal Symptom Rating Scale (GSRS) will be used to assess gastrointestinal function. The score ranges from 0-45. The higher score means poorer gastrointestinal function.
Quality of health and functional status | Before surgery and at the postoperative 3 months
  SF-36 consists of 36 items and is a short questionnaire to evaluate the health and functional status within one month. There are 8 dimensions regarding physiological functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. For each item, the average is 50 points, 0 is the lowest and 100 is the highest. The conversion score for each item is (the exact score minus the suspected lowest score) / (the difference between the expected highest and lowest score) × 100. The total score of the 8 dimensions is the total score of the scale.
Brain function | Before surgery and at the postoperative 3 months
  Resting functional magnetic resonance imaging (rs-fMRI) will measure brain structure and functional changes, including gray matter volume, gray matter thickness, functional connectivity.

IPD SHARING:
Plan to Share IPD: No